CLINICAL TRIAL: NCT02724748
Title: The Effectiveness of User-driven Intervention to Manage Patient Aggression in Mental Health Services
Brief Title: Managing Patient Aggression in Mental Health Services
Acronym: Violin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Academy of Finland (Other); Turku University Hospital (Other Government); Harvard Medical School (HMS and HSDM) (Other); Harvard School of Public Health (HSPH) (Other); Stanford University (Other); Sichuan University of China, China (Unknown); University of Nottingham (Other); World Health Organisation, Philippines (Unknown); The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Maritta Välimäki, Professor, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 294298
Record Dates: First submitted 2016-03-18; First posted 2016-03-31 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Aggression; Mental Disorders
Keywords: Aggression; Mental Health; Education, Continuing
MeSH Terms: conditions — Aggression; Mental Disorders; Psychological Well-Being | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational intervention (Experimental): Beside usual care the intervention will encourage collaborative practices between staff, patients and family members to adopt more human patient-centred approach on the unit. The intervention is designed to impact on treatment culture and thereby treatment practices on the study wards.
  Interventions: Behavioral: Educational intervention
- Treatment as usual (No Intervention): Wards allocated to comparison wards continue with their usual care. No restrictions on how nursing staff works in these wards, although participation in corresponding projects is not supported.

INTERVENTIONS:
Behavioral: Educational intervention — Educational intervention for staff members will encourage collaboration between patients, relatives and staff members. Skills, intellectual resources, motivation and encouragement among staff members to make changes on the unit will be supported. More detailed content of the intervention to be used in each unit will be tailored based on preparatory phase of the study and individual needs of the unit. The educational intervention will be carried out beside usual care.
  Arms: Educational intervention

SUMMARY:
To compare the effects of an educational intervention to usual practice (no specified staff education) on improving treatment culture and supporting team climate in staff members, which further could reduce the need for the use of coercive methods in psychiatric care.

DETAILED DESCRIPTION:
This is a single-blind, two-arm, cluster randomised controlled trial involving 28 psychiatric hospital wards across Finland.

Units are randomised on an equal basis to receive either staff educational programme (designed together with staff members, patients and relatives on the study units) or standard care. Inpatient psychiatric hospital organisations are the unit of randomisation. The cluster design will be used to avoid contamination between individual staff members in each study ward. We will use centralized randomisation at the University of Turku (Department of Mathematics and Statistics). Randomisation will be fully concealed and computer-generated by an independent statistician, who is not involved in the study. Investigators enrolling wards cannot foresee assignment. Outcome assessors and statisticians will be kept blinded to allocation. However, due to the type of intervention, allocation will be unmasked to patients and their relatives, contact persons in each ward, and health care staff delivering patient care on the wards after randomisation; this would reflect real-world care. While the Data Monitoring Committee undertook ongoing safety surveillance, investigators running the preliminary analysis for the Data Monitoring Committee will be masked to data until investigators released the database. Further, the statisticians and the National Register holder who are responsible in Finnish routine data used in this study, will be masked to ward allocation and patient data in each group. Randomisation will be done after collecting the baseline data from each unit.

Baseline data on coercive practices used on the units will be collected by the members of the research team with a help of staff members within the eight weeks, while observational and interview data related to the quality of the services will be collected by the research team (only in the intervention units). On the individual level, all staff members working in the study units, patients, and their relatives are eligible to participate in the study. Staff survey and interviews with staff members, patient groups and relatives will be done on the basis of free will. The staff of the unit/research team members will approach patients and their relatives to explain the purpose of the study and its arrangements orally and in written format. The opportunity to ask questions about the study will be given to them. Those that will be assessed having a lack of capacity to give informed consent and declined to participate will not be interviewed. Staff surveys will be repeated for baseline and follow-up. On the organisational level, the outcomes related to patient service use will be assessed 12 and 24 months after baseline data collection.

Assessing quality components: The strengths, weaknesses, opportunities, and threats related to the new practices will also be discussed and categorised based on SWOT analysis (Strength, Weakness, Opportunity, Threat). Possible barriers and facilitating factors for change on the on each unit will be identified. The quality of the service facilities will be assessed by observations on the units, based on World Health Organization's (2012) QualityRight Tool Kit focusing on five central quality criteria.

We have systematically searched for, but found no directly relevant past work. We assume that if the data will be obtained from local hospital registers by sampling 7 clusters (hospitals) with 265 subjects each in intervention group and 7 clusters with 265 subjects each in control group, we will have 80% power to detect a difference between the group proportions of -0.0400. The control group proportion is 0.1100. The intervention group proportion is assumed to be 0.1100 under the null hypothesis and 0.0700 under the alternative hypothesis. The test statistic used is the two-sided Z test (unpooled) with an overall significance level at 0.05. We may assume based on the hospital registers that sample size for the total population admitted in the study wards in one year will be 3710. However, if we consider a loss of 20% patients in the local care registers, the total number of patients on the randomised wards should be about 4454 patients. Further, if we assume 50% response rate for patient survey out of possible 3710 participants, we will assume that we will obtain 928 filled questionnaires during 6 month survey data collection period. The sample size calculation was adjusted for intra-cluster correlation at 0.005.

ELIGIBILITY:
Inclusion Criteria:

* Finnish speaking hospital organisations
* at least 1 psychiatric ward
* open 24/7
* are able to use coersive measures (seclusion room, limb restraint, forced medication, physical restraint)

Exclusion Criteria:

* wards specialised in forensic, psychogeriatric, or child and adolescent care alone
* similar type of project is underway or is planned to start

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of seclusion room use. | Three years
  The incidence of seclusion room use by patients in each unit.

SECONDARY OUTCOMES:
Other types of coercive measures | Three years
  Organisational outcomes. Incidence of other types of coercive measures used on patients (limb restraint, forced injection, physical restraint).
Service use | Three years
  Organisational outcomes. Type of admission, length of stay, deaths.
Team climate | 18-20 months after beginning of the intervention
  Staff outcomes. Team Climate Inventory, TCI.
Turnover | Three years
  Staff outcomes.
The functional capacity of patients | Nine months after beginning of the intervention
  Patient outcomes. Gobal Assessment Scale, GAS.
Patient treatment satisfaction | Nine months after beginning of the intervention
  Patient outcomes. Client Satisfaction Questionnaire, CSQ-8.
Quality of Life | Nine months after beginning of the intervention
  Patient outcomes. Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form, Q-LES-Q-SF

CONTACTS AND LOCATIONS:
Overall Officials: Maritta Välimäki, Professor, Study Director — University of Turku, Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valimaki M, Yang M, Normand SL, Lorig KR, Anttila M, Lantta T, Pekurinen V, Adams CE. Study protocol for a cluster randomised controlled trial to assess the effectiveness of user-driven intervention to prevent aggressive events in psychiatric services. BMC Psychiatry. 2017 Apr 4;17(1):123. doi: 10.1186/s12888-017-1266-6. PMID 28372555
- [Result] Valimaki M, Yang M, Vahlberg T, Lantta T, Pekurinen V, Anttila M, Normand SL. Trends in the use of coercive measures in Finnish psychiatric hospitals: a register analysis of the past two decades. BMC Psychiatry. 2019 Jul 26;19(1):230. doi: 10.1186/s12888-019-2200-x. PMID 31349787
- [Derived] Valimaki M, Lantta T, Anttila M, Vahlberg T, Normand SL, Yang M. An Evidence-Based Educational Intervention for Reducing Coercive Measures in Psychiatric Hospitals: A Randomized Clinical Trial. JAMA Netw Open. 2022 Aug 1;5(8):e2229076. doi: 10.1001/jamanetworkopen.2022.29076. PMID 36040740
- [Derived] Gibbon S, Khalifa NR, Cheung NH, Vollm BA, McCarthy L. Psychological interventions for antisocial personality disorder. Cochrane Database Syst Rev. 2020 Sep 3;9(9):CD007668. doi: 10.1002/14651858.CD007668.pub3. PMID 32880104
- See also: Study protocol — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5379524/pdf/12888_2017_Article_1266.pdf
- See also: Trends — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6660969/